CLINICAL TRIAL: NCT03278704
Title: Effects of Concurrent Resistance Exercise and High-intensity Interval Exercise Training on Skeletal Muscle Adaptations in Individuals With Type 2 Diabetes Mellitus
Brief Title: Concurrent Training in Type 2 Diabetes
Acronym: CONTRADIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment goal not met in allotted recruitment period
Sponsor: University of Birmingham (Other)
Collaborators: Loughborough University (Other); Metabolic Fitness Association, Italy (Other); Università degli studi di Roma Foro Italico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RG_16-218; ERN_16-1612 (Other: University of Birmingham ethics number); RRK6071 (Other: NHS R&D reference number)
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Concurrent training; Type 2 Diabetes Mellitus; Resistance exercise; High-Intensity Interval Training (HIIT); Muscle hypertrophy; Interference effect
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an exploratory randomized controlled trial. Participants will complete a parallel designed study, in which they will be randomly assigned to a resistance exercise (RE) only or concurrent RE and high-intensity interval training (RE + HIIT) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RE training only (Other): RE only - Progressive resistance exercise training only (leg extension, leg step up, chest press and pull down).
  Interventions: Other: RE only
- Concurrent RE + HIIT (Experimental): RE + HIIT - Progressive resistance exercise training (leg extension, leg step up, chest press and pull down) followed by HIIT (10 x 1 min at 90% heart rate maximum).
  Interventions: Other: RE + HIIT

INTERVENTIONS:
Other: RE only — 8 weeks of supervised training. Three times weekly with no more than two non-consecutive days without exercise.
  Arms: RE training only
Other: RE + HIIT — 8 weeks of supervised training. Three times weekly with no more than two non-consecutive days without exercise. Concurrent training: RE followed by HIIT within the same session.
  Arms: Concurrent RE + HIIT

SUMMARY:
It is recommended that individuals perform a combination of resistance exercise (RE) and endurance exercise. Lack of time is often cited as a reason for being unable to meet current exercise guidelines. Therefore, combining both forms in one session may be beneficial. However, research continues to elucidate whether interference of adaptive outcomes occurs when RE and endurance exercise are performed concurrently. A proposed interference effect suggests that concurrent training may dampen RE-induced adaptations (e.g., muscle strength and growth) compared to RE only.

The propose of this investigation is to determine the effects of concurrent RE and high-intensity interval training (HIIT), compared to RE only, on muscle health and cardiovascular risk in sedentary, middle-aged (40-65 years) who are overweight/obese with type 2 diabetes mellitus (T2DM). The investigators will measure the effects on muscle strength, muscle growth, cardiovascular fitness, glycaemic control and markers of cardiovascular risk before and after an 8-week training program. Data will be obtained through the analysis of skeletal muscle samples, blood samples, magnetic resonance imaging, questionnaires and exercise performance tests.It is hypothesized that concurrent RE + HIIT will amplify the exercise-induced muscle growth response, which will result in greater satellite cell content, compared to RE alone. As a result, this will lead to greater skeletal muscle mass and strength after RE + HIIT compared to RE in isolation.

A finding that concurrent resistance training and HIIT does not impede muscle adaptations could offer future strategies to minimize exercise time commitment whilst still maximizing the physiological benefits of both resistance and endurance exercise through a single training session. This may therefore provide an effective exercise strategy in the prevention and/or treatment of T2DM.

DETAILED DESCRIPTION:
Data analysis will be performed using IBM SPSS statistical software (IBM Corp., Armonk, New York, USA). All data will be checked for normality and appropriate log transformations applied prior to analysis of variance (ANOVA) for primary and secondary outcomes. Satellite cell content will be compared using a two-way, mixed-model ANOVA with one within (2 levels; pre- and post-training) and one between factor (2 level; exercise group) with significance set at P < 0.05.

Based on a mixed ANOVA with between- and within-participant factors, and previously published data (Babcock et al. 2012), a sample size of 24 participants (12 per group) will provide a power of 84%. This sample size will allow detection of a mean change in satellite cell content of 2.35, assuming standard deviations of the change from pre- to post-training as 2.266 and 1.331 in the two exercise groups. Sample size calculation was performed with an alpha error of 0.05. SamplePower 2.0 (SPSS Inc., Chicago, Illinois, USA) software was used to determine sample size.

This study will combine data collected at the University of Birmingham with previously collected data from an identical study design performed by a co-investigator (Dr Pugh) in Rome, Italy. The previous study has collected data from 10 participants across both exercise groups (RE, N = 7; RE + HIIT, N = 3). Therefore, it is necessary for the present study to recruit a further 14 participants (RE, N = 5, RE + HIIT, N = 9) in order to achieve a sample size of 24 participants (12 per group). However, based on an assumption of a 25% drop-out rate, the total minimal sample necessary will be 19 participants (RE, N = 7; RE + HIIT, N = 12).

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* White British/European
* Aged between 40 and 65 years at the time of screening
* Have a body mass index (BMI; body weight/height in m2) between 27 and 40 kg/m2
* Sedentary/untrained for at least 1 year (based on physical activity self-reports of fewer than two sessions of structured exercise per week last <30 min)
* T2DM (American Diabetes Association 2014) for more than 1 year
* Central obesity (defined as waist circumference ≥94 cm for males)

Exclusion Criteria:

* Currently involved in research or have recently (<6 months) been involved in any research prior to recruitment
* Any condition limiting or contraindicating physical activity; including diabetic peripheral neuropathy, and coronary or peripheral artery disease
* Previous myocardial infarction, previous or current angina, shortness of breath, or other symptoms suggestive of heart failure
* Insulin medication
* HbA1c more than 75 mmol/mol (9%)
* Uncontrollable hypertension: systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥100 mmHg
* Not weight stable for the last three months
* Smokers (within the last 12 months)
* Anticoagulant medication, such as warfarin or newer anticoagulant drugs. If participants are on aspirin medication, this would need to be stopped for 3 days prior to and during the day of any biopsy visit unless contraindicated (in which case participants would be excluded).

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Change in fibre-type specific satellite cell content | Prior to the 8-week training intervention and 72 hours after the last training session
  Assessed using immunofluorescence microscopy (Pax7-positive cells)

SECONDARY OUTCOMES:
Change in muscle-specific gene expression related to growth adaptations | Prior to the 8-week training intervention and 72 hours after the last training session
  Assessed using reverse-transcription polymerase chain reactions
Change in muscle fibre size | Prior to the 8-week training intervention and 72 hours after the last training session
  Assessed using immunofluorescence microscopy techniques to determine muscle fibre type-specific cross-sectional area
Change in muscle size | Prior to the 8-week training intervention and 48 hours after the last training session
  Assessed using MRI to determine whole and individual muscle group cross-section area and total muscle volume
Change in isometric muscle strength | Prior to the 8-week training intervention and 6 days after the last training session
  Assessed using a dynamometer
Change in isokinetic muscle strength | Prior to the 8-week training intervention and 6 days after the last training session
  Assessed using a dynamometer
Change in cardiorespiratory fitness | Prior to the 8-week training intervention and 6 days after the last training session
  Assessed using a V̇O2 peak test on a cycle ergometer
Change in habitual physical activity levels | Prior to the 8-week training intervention and 1 week after the last training session
  Assessed using 7-day continuous accelerometry data
Change in exercise enjoyment | After the first and last training session
  Assessed using validated questionnaires (PACES)
Change in glycaemic control | Prior to the 8-week training intervention and 72 hours after the last training session
  Assessed using blood analysis

CONTACTS AND LOCATIONS:
Overall Officials: Professor M Nimmo, PhD, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport, Exercise and Rehabilitation Sciences, University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] Babcock L, Escano M, D'Lugos A, Todd K, Murach K, Luden N. Concurrent aerobic exercise interferes with the satellite cell response to acute resistance exercise. Am J Physiol Regul Integr Comp Physiol. 2012 Jun 15;302(12):R1458-65. doi: 10.1152/ajpregu.00035.2012. Epub 2012 Apr 4. PMID 22492813